CLINICAL TRIAL: NCT03248206
Title: Effects of a Home-based Proprioceptive Neuromuscular Facilitation in Conjunction With Tendon Gliding Exercises on Sensorimotor Function in Upper Extremity of Subjects With Type 2 Diabetes Mellitus
Brief Title: Home-based Proprioceptive Neuromuscular Facilitation for Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-ER-105-257
Record Dates: First submitted 2017-08-07; First posted 2017-08-14 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2018-12

CONDITIONS: Diabetes Mellitus; Exercise
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF exercise program group (Active Comparator): The PNF home-program exercise group: perform grade 1&2 two times a day, at least 3 times per week, for 3 sets of 12 repetitions to increase neuromuscular and musculoskeletal endurance. (Grade 1: The participants performs the diagonal- spiral pattern that will enhance the strength or movement of a targeted muscle or muscle group.; Grade 2:The participants performs PNF exercise with elastic bands . )
  Interventions: Behavioral: lifestyle changes
- PNF in conjunction with tendon gliding exercise group (Experimental): Patients in PNF in conjunction with TGE group will perform PNF grade 1&2 as well as tendon gliding exercise two times a day, at least 3 times per week, for 3 sets of 10 repetitions. Training duration for both the two groups is twelve weeks.
  Interventions: Behavioral: lifestyle changes

INTERVENTIONS:
Behavioral: lifestyle changes — Providing a home-based exercise program supervised by therapists can be an acceptable strategy with the characteristics of convenience and inexpensiveness to promote neuromuscular and functional component for the patients with diabetes mellitus.

SUMMARY:
In this research work, the concept of strengthening technique of proprioceptive neuromuscular facilitation (PNF) incorporated with tendon gliding exercise (TGE) will be used to improve neuromuscular function of upper extremity of patients with diabetes mellitus. The first specific aim of the study is to examine the effects of home-based PNF exercise on the motor, sensation and functional performance parameters of upper extremity of the patients with diabetes mellitus. In addition, whether adding a tendon gliding exercise (TGE) to the home-based PNF exercises can provide better treatment effects for the patients with diabetes mellitus will also been investigated in this study. One of the hypothesis of this study is the prescribing home-based PNF exercise program has a positive treatment effect on neuromuscular function of the upper extremity of patients with diabetes mellitus. And,the other is home-based PNF in conjunction with TGE provides better benefits for neuromuscular function of the upper extremity of patients with diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Study participants will include clinically defined diabetic patients who are diagnosed based on the 1997 criteria of the American Diabetes Association. The inclusion criteria of the enrolled subjects are who suffered from neuropathy as diagnosed by abnormalities in either a nerve conduction study and / or quantitative sensory testing.

Exclusion Criteria:

* DM patients with (1) traumatic nerve injuries of the upper limbs, (2) trauma to the hand or congenital anomalies of the wrist and hand, (3) skin infections or disease, (4) known vascular complications of diabetes, such as stroke may have compromised the physical integrity of the patient, (5) grade 2 or higher arterial hypertension (>160/100 mmHg) or (6) cognitive deficits

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline result of Semmes-Weinstein monofilament (SWM) test at 12 weeks | pre-intervention (week 0), post-intervention (week 12) and follow-up evaluation (week 24)
  determine the touch-pressure threshold of the hands
Change from baseline result of Nerve conduction study (NCS) at 12 weeks | pre-intervention (week 0) and follow-up evaluation (week 24)
  determine nerve condition through detection of the amplitude of the sensory and motor nerve action potential
Change from baseline result of pinch-holding-up activity test at 12 weeks | pre-intervention (week 0), post-intervention (week 12) and follow-up evaluation (week 24)
  sensorimotor control of a hand
Change from baseline result of Purdue pegboard test at 12 weeks | pre-intervention (week 0), post-intervention (week 12) and follow-up evaluation (week 24)
  determine fine fingertip dexterity
Change from baseline result of Minnesota Manual Dexterity Test at 12 weeks | pre-intervention (week 0), post-intervention (week 12) and follow-up evaluation (week 24)
  determine unilateral and bilateral gross motor coordination of upper extremity
Change from baseline result of Manual tactile test at 12 weeks | pre-intervention (week 0), post-intervention (week 12) and follow-up evaluation (week 24)
  determine active touching sensation

SECONDARY OUTCOMES:
Change from baseline result of Grasp and pinch power at 12 weeks | pre-intervention (week 0), post-intervention (week 12) and follow-up evaluation (week 24)
  Grip strength of the hands will be assessed with a Jamar dynamometer
Change from baseline result of pinch power at 12 weeks | pre-intervention (week 0), post-intervention (week 12) and follow-up evaluation (week 24)
  Pinch power is measured with a pinch gauge
Change from baseline result of of shoulder flexion assessing by Micro FET hand-held dynamometer at 12 weeks | pre-intervention (week 0), post-intervention (week 12) and follow-up evaluation (week 24)
  Peak force of shoulder flexion (N) will be measured
Change from baseline result of shoulder internal rotation assessing by Micro FET hand-held dynamometer at 12 weeks | pre-intervention (week 0), post-intervention (week 12) and follow-up evaluation (week 24)
  Peak force of shoulder internal rotation (N) will be measured
Change from baseline result of shoulder external rotation assessing by Micro FET hand-held dynamometer at 12 weeks | pre-intervention (week 0), post-intervention (week 12) and follow-up evaluation (week 24)
  Peak force of shoulder external rotation (N) will be measured
Change from baseline result of peak torque of shoulder external rotation assessing by Bi-planar isokinetic dynamometer (BID) at 12 weeks | pre-intervention (week 0), post-intervention (week 12) and follow-up evaluation (week 24)
  Peak torque of shoulder external rotation (N⋅m) will be obtained
Change from baseline result of peak torque of shoulder internal rotation assessing by Bi-planar isokinetic dynamometer (BID) at 12 weeks | pre-intervention (week 0), post-intervention (week 12) and follow-up evaluation (week 24)
  Peak torque (PT) of shoulder internal rotation (N⋅m) will be obtained

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan